CLINICAL TRIAL: NCT05870891
Title: Equivalent Glycemic Load and Insulinemic Response Elicited by 7 Low Carbohydrate Products in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Mills (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INQ-2324
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy Nutrition
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Peanut Butter Cereal (Experimental): Consumption of Peanut Butter Cereal
  Interventions: Other: Food
- Cinnamon Almond Cereal (Experimental): Consumption of Cinnamon Almond Cereal
  Interventions: Other: Food
- Sriracha Crisps (Experimental): Consumption of Sriracha Crisps
  Interventions: Other: Food
- Cheddar Crisps (Experimental): Consumption of Cheddar Crisps
  Interventions: Other: Food
- Almond Blueberry Butter Bar (Experimental): Consumption of Almond Blueberry Butter Bar
  Interventions: Other: Food
- Peanut Butter and Dark Chocolate Bar (Experimental): Consumption of Peanut Butter and Dark Chocolate Bar
  Interventions: Other: Food
- Almond Dark Chocolate Bar (Experimental): Consumption of Almond Dark Chocolate Bar
  Interventions: Other: Food
- White Bread 5 g available carbohydrate (Experimental): Consumption of white bread containing 5 g available carbohydrate
  Interventions: Other: Food
- White Bread 20 g available carbohydrate (Active Comparator): Consumption of white bread containing 20 g available carbohydrate
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Food

SUMMARY:
The purpose of this study is to test the hypothesis that the equivalent glycemic load (EGL) value of portions of white bread containing 5 g available carbohydrate measured in this study is accurate and precise to within 1 gram. Additionally, the EGL of 7 low carbohydrate foods will be measured to determine their glycemic impact.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 inclusive
* Willing to abstain from unusual strenuous exercise and consuming alcoholic drinks for 24 hours before study days
* Willing to refrain from smoking tobacco or marijuana for 12h before and during study visits
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator
* Subjects must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria at screening
* Pregnant or lactating individuals
* Personal history of diabetes
* Major trauma or surgical event within 3 months of screening
* The presence of any laboratory result, health condition, illness or drug use that increases risk to the subject or to others or may affect the results, as judged by the Qualified Investigator
* Unwillingness or inability to comply with experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test meals. All allergens should be assumed to be a result of manufacturing practices.
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement or lifestyle modification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Equivalent glycemic load | -5 minutes to 120 minutes
  Equivalent glycemic load (EGL) for each test food, expressed as [EGL = T/(W/Cwb)] where T is the plasma glucose incremental area under the curve over 120 minutes (iAUC) elicited by one serving of test food, W is the mean iAUC elicited by the mean of two WB20 tests and Cwb is the amount of available carbohydrate in the WB20.

SECONDARY OUTCOMES:
Insulin iAUC over 120 minutes | -5 minutes to 120 minutes
  Postprandial serum insulin incremental area under the curve over 120 minutes for each food in a subset of n=10 individuals. Blood will be collected at -5, 0, 15, 30, 45, 60, 90, and 120 minutes.
Glucose iAUC over 120 minutes | -5 minutes to 120 minutes
  Postprandial plasma glucose incremental area under the curve over 120 minutes for each food in n=25 individuals. Blood will be collected at -5, 0, 15, 30, 45, 60, 90, and 120 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- INQUIS Clinical Research, Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data pertaining to glucose and insulin measurements will be shared upon reasonable request.
Time Frame: De-identified participant data pertaining to glucose and insulin measurements will be available after publication and will be available until 3 years after the publication date.
Access Criteria: Please contact the study sponsor to request access to the data.

REFERENCES:
- [Derived] Wolever TM, Miller K, Banh T. Equivalent Glycemic Load and Insulinemic Responses Elicited by Low-Carbohydrate Foods: A Randomized Trial in Healthy Adults. Curr Dev Nutr. 2025 Oct 30;9(12):107594. doi: 10.1016/j.cdnut.2025.107594. eCollection 2025 Dec. PMID 41439105